CLINICAL TRIAL: NCT06173336
Title: A Randomized Controlled Prospective Trial Comparing Clinical Outcomes and Efficacy of Single vs. Double Pyloromyotomy Technique for Gastric Peroral Endoscopic Pyloromyotomy (G-POEM) in the Treatment of Gastroparesis
Brief Title: Comparison of Outcomes for Single vs Double Pyloromyotomy for Gastroparesis Randomized Controlled Trial
Acronym: COMET-GP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 275425
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-09

CONDITIONS: Gastroparesis
Keywords: Gastric Per-Oral Endoscopic Myotomy (G-POEM)
MeSH Terms: conditions — Gastroparesis | interventions — Pyloromyotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single pyloromyotomy gastric per-oral endoscopic myotomy (G-POEM) (Active Comparator): Single cut pyloromyotomy technique during gastric per-oral endoscopic myotomy (G-POEM) procedure
  Interventions: Procedure: gastric per-oral endoscopic myotomy (G-POEM)
- Double pyloromyotomy gastric per-oral endoscopic myotomy (G-POEM) (Active Comparator): Double cut pyloromyotomy technique during gastric per-oral endoscopic myotomy (G-POEM) procedure
  Interventions: Procedure: gastric per-oral endoscopic myotomy (G-POEM)

INTERVENTIONS:
Procedure: gastric per-oral endoscopic myotomy (G-POEM) — Comparing single versus double pyloromyotomy in G-POEM for refractory and severe gastroparesis.

SUMMARY:
Gastroparesis is a chronic disease of the stomach that causes delayed gastric emptying without stenosis. The clinical symptoms of gastroparesis include nausea, vomiting, early satiety, post-prandial fullness, bloating, belching, and upper abdominal discomfort Gastroparesis cardinal symptoms index (GCSI) is a reliable, reproducible, and valid instrument for measuring symptom severity in patients with gastroparesis.

This will be a randomized controlled trial of all the patients who are referred to the University of Arkansas Medical Sciences (UAMS) for gastric peroral endoscopic pyloromyotomy (G-POEM) for treatment of refractory and severe gastroparesis. During G-POEM procedure, either single or double pyloromyotomy will be performed with randomization. The aim is to compare clinical outcomes and the efficacy of single versus double pyloromyotomy in G-POEM for refractory and severe gastroparesis.

DETAILED DESCRIPTION:
Gastroparesis is a chronic disease of the stomach that causes delayed gastric emptying without stenosis. It is a chronic alteration of gastric motility that leads to a delay in stomach emptying. It is an underdiagnosed condition. The prevalence is estimated at around 3% in the United States (mean age of 37.7 years, with an F: M ratio of 4:1. It is mainly an idiopathic condition; however, it can also be caused by diabetes mellitus and post-surgical conditions, such as fundoplication, vagotomy, bariatric surgery, and esophagectomy. Less frequently by conditions like post-infectious gastro-paresis, neurological or autoimmune diseases. The clinical symptoms of gastroparesis include nausea, vomiting, early satiety, post-prandial fullness, bloating, belching, and upper abdominal discomfort. The gastroparesis cardinal symptoms index (GCSI) is a reliable, reproducible, and valid instrument for measuring symptom severity in patients with gastroparesis. It is based on three sub-scales (post-prandial fullness/early satiety-4 items; nausea/vomiting-3 items; bloating-2 items), and each item ranges from 0 (none) to 5 (severe). GCSI is not a diagnostic tool, but it is helpful to measure the severity of the disease and the post-treatment improvement. Though the prevalence of gastroparesis has significantly increased over the last decade, management is still challenging. Patients with mild symptoms can be referred for dietary modifications coupled with medical therapy with prokinetics, especially metoclopramide. However, the response to prokinetics decreases over time. Moreover, these drugs have side effects, such as extrapyramidal symptoms and amenorrhea. Surgical approaches have been proposed; however, the invasive nature of those procedures and the low rate of clinical success have made them less favorable. Endoscopic interventions have also been described, including intra-pyloric injection of botulinum toxin, endoscopic gastrojejunostomy, and transpyloric stenting. For patients with refractory (persistent symptoms for >6 months refractory to medical therapy) and severe gastroparesis based on GCSI > 2, gastric per-oral endoscopic myotomy can be considered. In 2013, the first human gastric per-oral endoscopic myotomy (G-POEM) was performed. It was inspired by the per-oral endoscopic myotomy technique, with a similar dissection method, that allows pyloromyotomy. The technical steps of G-POEM involve mucosal incision about 5 cm from the pylorus with the creation of access to the submucosal plane after detaching the planes by injection of lifting solution; creation of the submucosal tunnel with dissection technique up to the duodenal bulb and exposure of the pylorus; verification of the integrity of the mucosal surface; pyloromyotomy and closure of the mucosal flap with multiple endoclips. In the single pyloromyotomy group, a selective circular pyloromyotomy is performed at the 6 or 7 o'clock position after identifying the pyloric ring. In the double pyloromyotomy group, another selective cut is performed at the 4 or 5 o'clock position to keep at least 1 cm between the two pyloromyotomies.

Only one retrospective case-controlled study compares single versus double pyloromyotomy at G-POEM for refractory gastroparesis. It showed a higher clinical response rate with double pyloromyotomy when compared with single pyloromyotomy in a 3- to 6-month follow-up period.

In this randomized controlled prospective multicenter study, the aim is to compare clinical outcomes and the efficacy of single versus double pyloromyotomy in G-POEM for refractory and severe gastroparesis. Prospective subjects will be approached regarding study inclusion either during a pre-endoscopy visit or shortly before the planned endoscopy procedure. If the latter, the prospective subject will be approached during intake and before being brought to the back for the procedure. The prospective subjects will be approached before any pre-procedure medication is administered. The study will be explained in detail and, if the prospective participant agrees, an informed consent form - HIPAA Research Authorization will be taken.

Prospective subjects will be randomized into one of two study groups: Single pyloromyotomy vs Double pyloromyotomy G-POEM using a computer-generated random sequence (prepared by the UAMS Biostatistics group) that will be placed in sealed envelopes. The envelopes will accompany the informed consent form will be opened after obtaining informed consent from the patients to determine their group assignment. The patient will open the envelop and hand it to the endoscopist performing the procedure.

Once randomized, the subjects will undergo the scheduled endoscopic procedure as planned.

Subjects will be followed up in the clinic at 3 months, 6 months, and 12 months (one year) after procedure per routine care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory (persistent symptoms for >6 months refractory to medical therapy) and severe gastroparesis based on GCSI > 2, with confirmed im-paired gastric emptying based on gastric emptying.
* Persons 18 years or older at the time of signing the informed consent

Exclusion Criteria:

* No previous attempt with at least one prokinetic drug.
* Previous gastric surgery.
* Esophageal or gastric varices and /or portal gastropathy.
* Pregnant patients.
* Malignant or pre-malignant gastric diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Clinical success at 3 months, 6 months and 12 months follow up | 3, 6 and 12 months
  Measuring clinical success
Gastroparesis Cardinal Symptom Index (GCSI) score before and after GPOEM at 3, 6 months and 12 months follow up | 3, 6 and 12 months
  Measuring GCSI scores
Technical success rate | At time of procedure
  Measuring technical success

SECONDARY OUTCOMES:
Total procedure time for each method | At time of procedure
  Documenting total time to perform procedure
Adverse events like pneumoperitoneum, gi bleeding, perforation, infection and abdominal pain | 0 and1 month
  Adverse events with both techniques
Recurrence of symptoms | 3, 6 and 12 months
  Any recurrence of gastroparesis symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sumant Inamdar, MD, Principal Investigator — University of Arkansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jung HK, Choung RS, Locke GR 3rd, Schleck CD, Zinsmeister AR, Szarka LA, Mullan B, Talley NJ. The incidence, prevalence, and outcomes of patients with gastroparesis in Olmsted County, Minnesota, from 1996 to 2006. Gastroenterology. 2009 Apr;136(4):1225-33. doi: 10.1053/j.gastro.2008.12.047. Epub 2008 Dec 24. PMID 19249393
- [Result] Verga MC, Mazza S, Azzolini F, Cereatti F, Conti CB, Drago A, Soro S, Elvo B, Grassia R. Gastric per-oral endoscopic myotomy: Indications, technique, results and comparison with surgical approach. World J Gastrointest Surg. 2022 Jan 27;14(1):12-23. doi: 10.4240/wjgs.v14.i1.12. PMID 35126859
- [Result] Camilleri M, Chedid V, Ford AC, Haruma K, Horowitz M, Jones KL, Low PA, Park SY, Parkman HP, Stanghellini V. Gastroparesis. Nat Rev Dis Primers. 2018 Nov 1;4(1):41. doi: 10.1038/s41572-018-0038-z. PMID 30385743
- [Result] Revicki DA, Rentz AM, Dubois D, Kahrilas P, Stanghellini V, Talley NJ, Tack J. Gastroparesis Cardinal Symptom Index (GCSI): development and validation of a patient reported assessment of severity of gastroparesis symptoms. Qual Life Res. 2004 May;13(4):833-44. doi: 10.1023/B:QURE.0000021689.86296.e4. PMID 15129893
- [Result] Lacy BE, Parkman HP, Camilleri M. Chronic nausea and vomiting: evaluation and treatment. Am J Gastroenterol. 2018 May;113(5):647-659. doi: 10.1038/s41395-018-0039-2. Epub 2018 Mar 15. PMID 29545633
- [Result] Hirsch W, Nee J, Ballou S, Petersen T, Friedlander D, Lee HN, Cheng V, Lembo A. Emergency Department Burden of Gastroparesis in the United States, 2006 to 2013. J Clin Gastroenterol. 2019 Feb;53(2):109-113. doi: 10.1097/MCG.0000000000000972. PMID 29256990
- [Result] Rao AS, Camilleri M. Review article: metoclopramide and tardive dyskinesia. Aliment Pharmacol Ther. 2010 Jan;31(1):11-9. doi: 10.1111/j.1365-2036.2009.04189.x. PMID 19886950
- [Result] Ahuja NK, Clarke JO. Pyloric Therapies for Gastroparesis. Curr Treat Options Gastroenterol. 2017 Mar;15(1):230-240. doi: 10.1007/s11938-017-0124-4. PMID 28124202
- [Result] Aghaie Meybodi M, Qumseya BJ, Shakoor D, Lobner K, Vosoughi K, Ichkhanian Y, Khashab MA. Efficacy and feasibility of G-POEM in management of patients with refractory gastroparesis: a systematic review and meta-analysis. Endosc Int Open. 2019 Mar;7(3):E322-E329. doi: 10.1055/a-0812-1458. Epub 2019 Feb 28. PMID 30842971
- [Result] Khashab MA, Stein E, Clarke JO, Saxena P, Kumbhari V, Chander Roland B, Kalloo AN, Stavropoulos S, Pasricha P, Inoue H. Gastric peroral endoscopic myotomy for refractory gastroparesis: first human endoscopic pyloromyotomy (with video). Gastrointest Endosc. 2013 Nov;78(5):764-8. doi: 10.1016/j.gie.2013.07.019. No abstract available. PMID 24120337
- [Result] Abdelfatah MM, Li B, Kapil N, Noll A, Li L, Luo H, Chen H, Xia L, Chen X, Patel V, Mekaroonkamol P, Massaad J, Keilin S, Cai Q. Short-term outcomes of double versus single pyloromyotomy at peroral endoscopic pyloromyotomy in the treatment of gastroparesis (with video). Gastrointest Endosc. 2020 Sep;92(3):603-609. doi: 10.1016/j.gie.2020.01.016. Epub 2020 Jan 17. PMID 31958460